CLINICAL TRIAL: NCT05708781
Title: Efficacy of Core Strengthening and Intensive Dynamic Back Exercises on Pain, Muscle Strength, Endurance, and Functional Disability in Patients With Chronic Non-specific Low Back Pain. a Randomized Comparative Study
Brief Title: Efficacy of Core Strengthening and Intensive Dynamic Back Exercises in Patient With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Najran University (Other)
Responsible Party: Principal Investigator, Hashim Ahmed, Assistant Professor, Najran University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IE/IIMS&R/2022/43
Record Dates: First submitted 2023-01-20; First posted 2023-02-01 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CSE Group (Experimental): in addition to Conventional treatment, core strengthening exercise were given
  Interventions: Other: Core strengthening exercise; Other: Control group
- IDBE Group (Experimental): in addition to Conventional treatment, intensive dynamic back exercise were given
  Interventions: Other: intensive dynamic back exercise; Other: Control group
- Control Group (Active Comparator): Conventional Treatment
  Interventions: Other: Control group

INTERVENTIONS:
Other: Core strengthening exercise — 1. Isolated lumbar stabilization muscle training:
  2. Bridge track:
  3. Dead bug track:
  4. Quadruped Track:
  5. Supine Track:
  6. Side-support Track:
  7. Prone Track:
  8. Standing Track:
  Arms: CSE Group
Other: intensive dynamic back exercise — 1. Trunk lifting Prone on a couch, hips at the edge, upper part of the body free but supported by the hands against the floor. Strap fixation over the calves. With hands on the forehead, the trunk is lifted to the greatest possible extension in hips and spine. If necessary, starting with support from physical therapist. During pauses a chair in front of the couch supports the patient.
  2. Leg lifting Standing by the end of the couch, leaning over to a prone position with the hips against the edge in 90 degree flexion, knees 45 degree and feet on the floor. Strap fixation over the chest. Straps around knees to keep legs together. Both legs are straightened and lifted to the greatest possible extension in hips and spine. Again support from physical therapist is necessary.
  3. Pull to neck Sitting on a tool with the arms straight and abducted over the head and hands grasping a weight lever. Against sub-maximal resistance the lever is pulled behind neck and shoulders.
  Arms: IDBE Group
Other: Control group — Hot Pack was given for twenty minutes, slow sustained stretching exercises ( 20 second hold, 10- second relaxation) were given, and isometric exercise of the back((10 repetitions of two sets with 10 seconds hold) alternate days for six weeks.

SUMMARY:
The study aimed to investigate the efficacy of core strengthening and intensive dynamic back exercises on pain, muscle strength, endurance, and functional disability in patients with chronic non-specific low back pain.

DETAILED DESCRIPTION:
The study will be based on a three-arm parallel group randomized control design. Forty-five participants with chronic non-specific low back pain will be recruited from the Physiotherapy department, at Integral University, India. Study objectives and procedure will be properly explained and written informed consent will be obtained at the beginning of the study. All the participants will be randomly divided into three groups A, B, and C. Experimental group A will be receiving the hot pack, active Stretching, isometric exercise intervention, and core strengthening exercises while group B will receive the hot pack, active Stretching, isometric exercise intervention, and intensive dynamic back exercises, control group C will receive the hot pack, active Stretching, isometric exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* age 20-50 years
* chronic low back pain (>3 months),

Exclusion Criteria:

* Participants with low back pain related to cancer,
* infection,
* inflammatory arthropathy,
* high-velocity trauma,
* fracture
* low back pain associated with severe or progressive neurological deficits trauma
* pregnancy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 6 Weeks
  The pain intensity was assessed Using a numeric pain rating scale (NPRS), It's a 11 point scale, where zero indicates no pain and 10 indicates severe pain
functional Limitation | 6 Weeks
  Functional limitation was assessed by using Oswestry disability Index questionnaire Each section is scored on a 0-5 scale, 5 representing the greatest disability.
Muscle Endurance | 6 Weeks
  Muscle endurance was assessed by using timed endurance tests including the extensor endurance test, flexor endurance test and the side bridge test. The hold time was recorded in seconds once the patient was not able to maintain the respective endurance test position.

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Ahmed, PhD, Principal Investigator — Najran University
Locations (2):
- Integral University Hospital, Lucknow, Uttar Pardesh, India
- Hashim Ahmed, Najrān, Najran Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No